CLINICAL TRIAL: NCT04411043
Title: Prospective and Retrospective Study Evaluating Epidemiological, Clinical, Molecular and Therapeutic Data of Prolymphocytic Leukemia T. A FILO Study.
Brief Title: Observatory of Prolymphocytic Leukemia T
Acronym: T-PLL
Status: Recruiting | Type: Observational
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: T-PLL
Record Dates: First submitted 2020-05-13; First posted 2020-06-02 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Prolymphocytic Leukemia; T-cell Leukemia
MeSH Terms: conditions — Leukemia, Prolymphocytic; Leukemia, T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — bone marrow and peripheral blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Molecular caracterization — Prospective and retrospective study evaluating the epidemiological, clinical, molecular and therapeutic data of prolymphocytic leukemias T

SUMMARY:
Prolymphocytic leukemia T is a rare disease representing approximately 2% of mature lymphoid leukemias and 20% of prolymphocytic leukemias. It mainly affects the elderly with an aggressive clinical course. It is a hemopathy exhibiting a post thymic T phenotype (Tdt-, CD1a-, CD5 +, CD2 + and CD7 +), generally CD4 + / CD8-, but also CD4 + / CD8 + or CD8 + / CD4-.

The main feature of T-PLL is the rearrangement of chromosome 14 involving genes encoding the T cell receptor complex (TCR) subunits, leading to overexpression of the proto-oncogene TCL1.

On the molecular level, the study of Prolymphocytic leukemia T shows a substantial mutational activation of the IL2RG-JAK1-JAK3-STAT5B axis.

Patients with Prolymphocytic leukemia T have a poor prognosis, due to a poor response to conventional chemotherapy. Treatment with the anti-CD52 monoclonal antibody: alemtuzumab has considerably improved the results, but the responses to treatment are transient; therefore, patients who obtain a response to alemtuzumab treatment are candidates for stem cell allograft (TSS) if they are eligible for this procedure. This combined approach extended the median survival to four years or more. However, new approaches using well-tolerated therapies that target signaling and survival pathways are necessary for most patients who are unable to receive intensive chemotherapy, such as JAK STAT axis inhibitors, anti-AKT, or anti BCL2 .

Main objective: Better manage prolymphocytic T leukemias.

Secondary objectives:

* Molecular characterization of prolymphocytic leukemia T.
* Study of the response to treatment, disease-free survival, overall survival.
* Impact of prognostic factors on response to treatment, and survival.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 or over
* Patient with prolymphocytic T leukemia

Exclusion Criteria:

* Absence of signature of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with prolymphocytic T leukemia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics of prolymphocytic leukemia T | from day 0 through study completion, an average of 3 years
  pathology description at diagnosis and its evolution over time
Biological characteristics of prolymphocytic leukemia T | At day 0 and at relapse, an average of 3 years
  Blood count : Hemoglobin, Leukocytes, Lymphocytes, Platelets, Eosinophils (giga / liters)
Flow cytometry data of bone marrow and blood cells | At day 0 and at relapse, an average of 3 years
  Positive or negative immunophenotyping
karyotype of tumor cells | At day 0 and at relapse, an average of 3 years
  karyotipic formula

CONTACTS AND LOCATIONS:
Overall Officials: Kamel LARIBI, Dr, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Chd Le Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: No